CLINICAL TRIAL: NCT06686602
Title: Assessing Risk Factors Associated With the Onset of Oral Mucositis/Stomatitis and Ocular Surface Events (OSE) in Patients With Non-small Cell Lung Cancer (NSCLC) and HER2-negative Breast Cancer (BC)
Brief Title: A Study Assessing Risk Factors for Oral Mucositis/Stomatitis and Ocular Surface Events in NSCLC and Breast Cancer
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS1062-0008-NIS-EPI
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Advanced/Metastatic NSCLC; Advanced/Metastatic HER2-negative Breast Cancer
Keywords: Advanced/metastatic non-small cell lung cancer (NSCLC); Advanced/metastatic human epidermal growth factor receptor 2 (HER2)-negative breast cancer; Oral mucositis/stomatitis; Ocular surface events
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSCLC: Adult patients diagnosed with advanced or metastatic (stage IIIB/IIIC or IV) non-small cell lung cancer (NSCLC).
  Interventions: Other: No drug
- HER2-negative Breast Cancer: Adult patients diagnosed with advanced or metastatic (stage IIIB/IIIC or IV) human epidermal growth factor receptor 2 (HER2)-negative breast cancer.
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — This is a non-interventional study and no study drug will be administered.

SUMMARY:
This study will identify risk factors for oral mucositis/stomatitis and ocular surface events (OSE) in patients with advanced/metastatic non-small cell lung cancer (NSCLC) and advanced/metastatic human epidermal growth factor receptor 2 (HER2)-negative breast cancer.

DETAILED DESCRIPTION:
It is important to identify risk factors for the onset of oral mucositis/stomatitis and OSE to identify high-risk patients who will be taking Dato-DXd. Understanding these risk factors in patients receiving standard-of-care anti-cancer therapies may also help with mitigation strategies. This objective will be achieved by identifying and describing patient demographics and clinical characteristics of cases with oral mucositis/stomatitis and OSE. No study drug will be provided or administered for this study.

ELIGIBILITY:
Inclusion Criteria

1. The inclusion criteria for the NSCLC cohort consists of patients with advanced or metastatic (stage IIIB/IIIC or IV) NSCLC diagnosis between January 1, 2015 and December 31, 2023 who are at least 18 years old at the time of first diagnosis (cohort entry date) and treated with at least one line of therapy (LOT) for advanced/metastatic disease.
2. The inclusion criteria for the breast cancer cohort consists of female patients with advanced or metastatic (stage IIIB/IIIC and IV) HER2-negative BC diagnosis between January 1, 2012 and December 31, 2023 who are at least 18 years old at the time of first diagnosis (cohort entry date) and treated with at least one LOT for advanced/metastatic disease.

Exclusion Criteria

1) The exclusion criteria for both cohorts consist of patients with other primary cancer type prior to the cohort entry date and patients who are pregnant 9 months (275 days) prior to, on, or after the cohort entry date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This nested case-control study is conducted in cohorts of adult patients diagnosed with advanced or metastatic (stage IIIB/IIIC, or IV) NSCLC and advanced or metastatic HER2-negative breast cancer. The time period is 2015 to 2023 for the NSCLC cohort and 2012 to 2023 for the breast cancer cohort. This time period was selected to account for the post-immunotherapy era for NSCLC and post-everolimus era for breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 13759 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Patient Demographics in NSCLC and Breast Cancer Patients With Oral Mucositis/Stomatitis or OSE Compared with Patients Without Oral Mucositis/Stomatitis or OSE | From NSCLC diagnosis (01 January 2015) or Breast Cancer diagnosis (01 January 2012) up to until death, exit from the database, or March 31, 2024, whichever comes first (approximately 12 years 2 months)
Clinical Characteristics in NSCLC and Breast Cancer Patients With Oral Mucositis/Stomatitis or OSE Compared with Patients Without Oral Mucositis/Stomatitis or OSE | From NSCLC diagnosis (01 January 2015) or Breast Cancer diagnosis (01 January 2012) up to until death, exit from the database, or March 31, 2024, whichever comes first (approximately 12 years 2 months)

CONTACTS AND LOCATIONS:
Locations (1):
- ConcertAI Database, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No